CLINICAL TRIAL: NCT03226275
Title: A Randomized, Two-period Crossover Trial Examining Bioequivalence of Bisoprolol-Amlodipine 5 mg/5 mg Combination Tablets Versus Bisoprolol 5 mg Tablets and Amlodipine 5 mg Tablets Given Concomitantly in Healthy Subjects in Fasting and Fed State
Brief Title: Bioequivalence Trial of Concor AM® vs Bisoprolol and Amlodipine in Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EMR200006-001
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: Concor AM®; Concor®; Norvasc®; Bisoprolol; Amlodipine; Bisoprolol-Amlodipine fixed dose combination; Chinese Participants
MeSH Terms: interventions — Bisoprolol; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fasting: First Bisoprolol-Amlodipine FDC, Then Both Separately (Experimental): Participants received a single oral dose of 5 milligram(mg)/5 mg bisoprolol-amlodipine FDC tablet (Concor AM®) on Day 1 in treatment period 1 followed by a single oral dose of 5 mg bisoprolol and a single oral dose of 5 mg amlodipine given concomitantly on Day 15 in treatment period 2 under fasting conditions. The two periods were separated by a washout period of 14 days.
  Interventions: Drug: Bisoprolol-Amlodipine FDC; Drug: Bisoprolol; Drug: Amlodipine
- Fasting: First Bisoprolol and Amlodipine Separately, Then FDC (Experimental): Participants received a single oral dose of 5 mg bisoprolol and a single oral dose of 5 mg amlodipine given concomitantly on Day 1 in treatment period 1 followed by a single oral dose of 5 mg/5 mg bisoprolol-amlodipine FDC tablet (Concor AM®) on Day 15 in treatment period 2 under fasting conditions. The two periods were separated by a washout period of 14 days.
  Interventions: Drug: Bisoprolol-Amlodipine FDC; Drug: Bisoprolol; Drug: Amlodipine
- Fed: First Bisoprolol-Amlodipine FDC, Then Both Separately (Experimental): Participants received a single oral dose of 5 mg/5 mg bisoprolol-amlodipine FDC tablet (Concor AM®) on Day 1 in treatment period 1 followed by a single oral dose of 5 mg bisoprolol and a single oral dose of 5 mg amlodipine given concomitantly on Day 15 in treatment period 2 under fed conditions. The two periods were separated by a washout period of 14 days.
  Interventions: Drug: Bisoprolol-Amlodipine FDC; Drug: Bisoprolol; Drug: Amlodipine
- Fed: First Bisoprolol and Amlodipine Separately, Then FDC (Experimental): Participants received a single oral dose of 5 mg bisoprolol and a single oral dose of 5 mg amlodipine given concomitantly on Day 1 in treatment period 1 followed by a single oral dose of 5 mg/5 mg bisoprolol-amlodipine FDC tablet (Concor AM®) on Day 15 in treatment period 2 under fed conditions. The two periods were separated by a washout period of 14 days.
  Interventions: Drug: Bisoprolol-Amlodipine FDC; Drug: Bisoprolol; Drug: Amlodipine

INTERVENTIONS:
Drug: Bisoprolol-Amlodipine FDC — Participants received a single oral dose of 5 milligram(mg)/5 mg bisoprolol-amlodipine FDC tablet (Concor AM®) either on Day 1 or Day 15 under fasting or fed conditions.
  Other Names: Concor AM®
Drug: Bisoprolol — Participants received 5 mg bisoprolol tablet as a single oral dose either on Day 1 or Day 15 under fasting or fed conditions.
Drug: Amlodipine — Participants received 5 mg amlodipine tablet as a single oral dose either on Day 1 or Day 15 under fasting or fed conditions.

SUMMARY:
This is a Phase I, open-label, randomized, 2-period, 2-sequence, crossover study to demonstrate bioequivalence (BE) between the bisoprolol-amlodipine fixed-dose-combination (FDC) tablet (investigational product) and bisoprolol and amlodipine tablets administered concomitantly (comparators) given as a single oral dose in fasting and fed state.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the entire trial period and willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer
* Chinese male and female volunteer
* Volunteer with a body mass index greater than or equal to 18 and below 28 kilogram/meter^2 (kg/m^2)
* Systolic blood pressure (in supine position) within 100 to 139 mmHg (inclusive) and diastolic blood pressure (in supine position) within 65 to 90 millimeter of mercury (mmHg) (inclusive) at Screening, during Admission to the Clinical Research Unit (CRU) (12 hour predose) and before each dosing
* Clinical laboratory values (within 1 month before screening) within the laboratory's stated normal range; if not within this range, they must lack clinical significance
* Healthy according to assessment of the medical history, Electrocardiogram, vital signs, physical examination,laboratory results, negative drug screening, and negative serology tests (except results after vaccination)
* Non-smoker or ex-smoker, not using any nicotine product; an ex-smoker being defined as someone who completely stopped smoking for at least 12 months before Day 1 of the trial
* Each participant has to be capable of understanding the trial procedures and sign the Informed consent form prior to their participation in the trial
* Participants must consent to adhere to the recommended contraceptive methods

Exclusion Criteria:

* Significant history of hypersensitivity to bisoprolol, amlodipine, other dihydropyridines, or any related products (including excipients of the formulations)
* Significant history of severe hypersensitivity reactions (eg, angioedema) to any drugs
* Pulse rate (in supine position) less than (<) 60 beats per minute (bpm) or more than 100 bpm at screening
* Presence of significant arrhythmia: QTc interval prolongation (QTc greater than 430 milliseconds (msec), severe sinus node dysfunction, or second or third atrioventricular block
* History of low blood pressure (< 100/65 mmHg) or vegetative dystonia
* History or presence of peripheral arterial occlusion or Raynaud's syndrome
* Presence of diabetes mellitus
* History or presence of asthma
* Presence of significant gastrointestinal, liver, kidney disease, surgery, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or known to potentiate or predispose to undesired effects
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, and human immunodeficiency virus [HIV] antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin, St. John's wort or other herbal medicine known with effect on CYP enzymes) within 28 days before Day 1 of this trial
* Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, endocrine, immunologic, or dermatological disease
* Presence or history of significant angina pectoris, acute myocardial infarction or ST segment and T wave changes other than non-clinically significant minor changes
* Presence or history of ventricular arrhythmia (such as ventricular tachycardia or ventricular fibrillation) or of congestive heart failure Acute conditions which might alter the renal function (eg, dehydration, severe infection)
* Surgery in the previous 28 days before Day 1 of this trial
* Any history of tuberculosis and/or prophylaxis for tuberculosis within 10 years of Day 1 of the trial
* Positive results to HIV antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or treponema pallidum (TP) antibody tests
* Donation of 50 milliliter (mL) or more of blood within 28 days before Day 1 of the trial; donation of 500 mL or more of blood within 56 days before Day 1 of the trial
* History of suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
* Poor motivation, intellectual problems likely to limit the validity of consent to participate in the trial or limit the ability to comply with the protocol requirements or inability to cooperate adequately, inability to understand and to observe the instructions of the physician
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 × 14 gram (g) alcohol per day, intake of excessive alcohol, acute or chronic use)
* Positive urine screening of drugs of abuse (cannabis, benzodiazepines, barbiturates, opiates, cocaine, and methyl amphetamine), or positive breath test of alcohol
* Positive pregnancy test (only for females of child-bearing potential) or females breast feeding a child
* Consumption of large quantities of methylxanthine-containing beverages (more than 600 mg caffeine/day: 1 cup (250 mL) of coffee contains approximately 100 mg of caffeine, 1 cup of black or green tea contains approximately 30 mg and 1 glass of cola contains approximately 20 mg caffeine)
* Volunteers who took an investigational product (in another clinical trial) by prescription within 2 weeks or an over-the-counter medication taken within 1 week before drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2017-09-09 (Actual); Study Completion 2017-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Xuanwu Hospital, Beijing, China

REFERENCES:
- [Derived] Hu C, Hu X, Wang C, Zhao Z, Gao D, Chen X, Zhou D, Huang Y, Li L, Zhang L. Bioequivalence and Pharmacokinetics of Bisoprolol-Amlodipine 5 mg/5 mg Combination Tablet versus Bisoprolol 5 mg Tablet and Amlodipine 5 mg Tablet: An Open-Label, Randomized, Two-Sequence Crossover Study in Healthy Chinese Subjects. Clin Drug Investig. 2018 Dec;38(12):1145-1154. doi: 10.1007/s40261-018-0700-y. PMID 30232699

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was designed to assess bioequivalence (BE) between a single oral dose of bisoprolol-amlodipine fixed-dose-combination (FDC) tablet and bisoprolol and amlodipine, each given concomitantly as a single dose in fasting or fed state.
Period: Treatment Period 1 (8 Days)
Arm/Group | Fasting: First Bisoprolol-Amlodipine FDC, Then Both Separately | Fasting: First Bisoprolol and Amlodipine Separately, Then FDC | Fed: First Bisoprolol-Amlodipine FDC, Then Both Separately | Fed: First Bisoprolol and Amlodipine Separately, Then FDC
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 1 | 1
Not completed — Did not pass blood pressure examination | 0 | 0 | 1 | 0
Not completed — Protocol non-compliance | 0 | 0 | 0 | 1
Period: Treatment Period 2 (8 Days)
Arm/Group | Fasting: First Bisoprolol-Amlodipine FDC, Then Both Separately | Fasting: First Bisoprolol and Amlodipine Separately, Then FDC | Fed: First Bisoprolol-Amlodipine FDC, Then Both Separately | Fed: First Bisoprolol and Amlodipine Separately, Then FDC
Started | 8 | 8 | 7 | 7
Completed | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasting: First Bisoprolol-Amlodipine FDC, Then Both Separately | Fasting: First Bisoprolol and Amlodipine Separately, Then FDC | Fed: First Bisoprolol-Amlodipine FDC, Then Both Separately | Fed: First Bisoprolol and Amlodipine Separately, Then FDC | Total
Number analyzed (Participants) | 8 | 8 | 7 | 7 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (8.89) | 29.3 (3.15) | 31.0 (3.56) | 32.4 (10.29) | 31.6 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 3 | 11
  Male | 4 | 6 | 5 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 7 | 7 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Bisoprolol and Amlodipine
Time Frame: Pre-dose (Baseline) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose for each treatment period
Population: The Pharmacokinetic (PK) Analysis Set included all participants who completed the study with adequate study medication compliance, without any relevant protocol violations with respect to factors likely to affect comparability of PK results, and with sufficient evaluable data to determine primary endpoints (AUC0-t and Cmax ) for both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Groups:
- Fasting: Bisoprolol-Amlodipine FDC: All participants who received a single oral dose of 5 mg/5 mg bisoprolol-amlodipine FDC tablet as a single oral dose on Day 1 or Day 15 under fasting conditions.
- Fasting: Bisoprolol and Amlodipine Separately: All participants who received a single dose of 5 mg bisoprolol and a single dose of 5 mg amlodipine given concomitantly on Day 1 or Day 15 under fasting conditions.
- Fed: Bisoprolol-Amlodipine FDC: All participants who received a single oral dose of 5 mg/5 mg bisoprolol-amlodipine FDC tablet as a single oral dose on Day 1 or Day 15 under fed conditions.
- Fed: Bisoprolol and Amlodipine Separately: All participants who received a single dose of 5 mg bisoprolol and a single dose of 5 mg amlodipine given concomitantly on Day 1 or Day 15 under fed conditions.
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
nanogram hour per milliliter (ng*h/mL)
  Bisoprolol | 294 (16.7) | 295 (21.5) | 270 (23.4) | 275 (23.9)
  Amlodipine | 205 (32.1) | 212 (34.7) | 174 (29.9) | 167 (33.5)
Statistical Analysis 1: Comparison: Fasting: Bisoprolol-Amlodipine FDC vs Fasting: Bisoprolol and Amlodipine Separately; Statistical Comparison of Bisoprolol in Fasting state; Test type: Equivalence — Results based on a mixed-effects model with sequence, treatment, and period as fixed effects and participant nested within sequence as a random effect; Geometric Least Square Mean Percentage = 99.46, 90% CI 2-sided [93.25 to 106.09]
Statistical Analysis 2: Comparison: Fasting: Bisoprolol-Amlodipine FDC vs Fasting: Bisoprolol and Amlodipine Separately; Statistical Comparison of Amlodipine in Fasting State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 96.76, 90% CI 2-sided [92.95 to 100.73]
Statistical Analysis 3: Comparison: Fed: Bisoprolol-Amlodipine FDC vs Fed: Bisoprolol and Amlodipine Separately; Statistical Comparison of Bisoprolol in Fed State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 98.95, 90% CI 2-sided [90.02 to 108.76]
Statistical Analysis 4: Comparison: Fed: Bisoprolol-Amlodipine FDC vs Fed: Bisoprolol and Amlodipine Separately; Statistical Comparison of Amlodipine in Fed State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 103.07, 90% CI 2-sided [95.53 to 111.20]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bisoprolol and Amlodipine
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
ng/mL
  Bisoprolol | 26.1 (20.1) | 26.6 (21.2) | 20.5 (18.6) | 21.9 (27.2)
  Amlodipine | 4.17 (25.6) | 4.17 (24.1) | 3.34 (23.1) | 3.19 (31.7)
Statistical Analysis 1: Comparison: Fasting: Bisoprolol-Amlodipine FDC vs Fasting: Bisoprolol and Amlodipine Separately; Statistical Comparison of Bisoprolol in Fasting State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 97.85, 90% CI 2-sided [92.29 to 103.74]
Statistical Analysis 2: Comparison: Fasting: Bisoprolol-Amlodipine FDC vs Fasting: Bisoprolol and Amlodipine Separately; Statistical Comparison of Amlodipine in Fasting State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 100.03, 90% CI 2-sided [94.37 to 106.03]
Statistical Analysis 3: Comparison: Fed: Bisoprolol-Amlodipine FDC vs Fed: Bisoprolol and Amlodipine Separately; Statistical Comparison of Bisoprolol in Fed State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 93.87, 90% CI 2-sided [84.56 to 104.20]
Statistical Analysis 4: Comparison: Fed: Bisoprolol-Amlodipine FDC vs Fed: Bisoprolol and Amlodipine Separately; Statistical Comparison of Amlodipine in Fed State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 106.56, 90% CI 2-sided [97.82 to 116.08]

3. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Bisoprolol and Amlodipine
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set.
Measure: Median (Full Range); unit: hours
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
hours
  Bisoprolol | 1.00 [1.00 to 3.00] | 1.00 [0.500 to 2.00] | 3.00 [1.00 to 6.00] | 3.00 [2.00 to 6.00]
  Amlodipine | 6.00 [4.00 to 8.00] | 6.00 [4.00 to 12.0] | 6.00 [4.00 to 15.0] | 6.00 [4.00 to 10.0]
Statistical Analysis 1: Comparison: Fasting: Bisoprolol-Amlodipine FDC vs Fasting: Bisoprolol and Amlodipine Separately; Statistical Comparison of Bisoprolol in Fasting State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Median Difference = 0.13, 90% CI 2-sided [0.00 to 0.50]
Statistical Analysis 2: Comparison: Fasting: Bisoprolol-Amlodipine FDC vs Fasting: Bisoprolol and Amlodipine Separately; Statistical Comparison of Amlodipine in Fasting State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Median Difference = 0.00, 90% CI 2-sided [-1.00 to 0.00]
Statistical Analysis 3: Comparison: Fed: Bisoprolol-Amlodipine FDC vs Fed: Bisoprolol and Amlodipine Separately; Statistical Comparison of Bisoprolol in Fed State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Median Difference = 0.00, 90% CI 2-sided [-1.00 to 0.50]
Statistical Analysis 4: Comparison: Fed: Bisoprolol-Amlodipine FDC vs Fed: Bisoprolol and Amlodipine Separately; Statistical Comparison of Amlodipine in Fed State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Median Difference = 0.00, 90% CI 2-sided [-1.00 to 0.50]

4. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Bisoprolol and Amlodipine
Description: Apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination. Terminal half-life was calculated as ln(2)/λz, where λz is a terminal rate constant, which was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set. Here, "Number Analyzed" signified those participants who were evaluable for the specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
hours
  Bisoprolol | 8.87 (18.1) | 8.84 (15.4) | 9.49 (30.2) | 8.86 (20.6)
  Amlodipine: number analyzed (Participants) | 15 | 13 | 13 | 14
  Amlodipine | 51.8 (16.1) | 49.7 (23.5) | 46.7 (16.5) | 43.2 (26.1)

5. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC 0-inf) of Bisoprolol and Amlodipine
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
ng*h/mL
  Bisoprolol | 306 (16.6) | 306 (21.5) | 281 (23.4) | 287 (23.2)
  Amlodipine: number analyzed (Participants) | 15 | 13 | 13 | 14
  Amlodipine | 235 (34.4) | 216 (31.7) | 192 (31.4) | 182 (34.8)
Statistical Analysis 1: Comparison: Fasting: Bisoprolol-Amlodipine FDC vs Fasting: Bisoprolol and Amlodipine Separately; Statistical Comparison of Bisoprolol in Fasting State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 99.98, 90% CI 2-sided [93.61 to 106.79]
Statistical Analysis 2: Comparison: Fasting: Bisoprolol-Amlodipine FDC vs Fasting: Bisoprolol and Amlodipine Separately; Statistical Comparison of Amlodipine in Fasting State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 98.68, 90% CI 2-sided [93.38 to 104.28]
Statistical Analysis 3: Comparison: Fed: Bisoprolol-Amlodipine FDC vs Fed: Bisoprolol and Amlodipine Separately; Statistical Comparison of Bisoprolol in Fed State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 98.52, 90% CI 2-sided [89.75 to 108.15]
Statistical Analysis 4: Comparison: Fed: Bisoprolol-Amlodipine FDC vs Fed: Bisoprolol and Amlodipine Separately; Statistical Comparison of Amlodipine in Fed State; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Percentage = 104.06, 90% CI 2-sided [96.11 to 112.66]

6. Secondary Outcome: Extrapolated Part of Area Under the Plasma Concentration Curve From Time Zero to Infinity (AUCextra%) of Bisoprolol and Amlodipine
Description: AUCextra% was calculated as area under the curve from time tlast extrapolated to infinity given as percentage of AUC 0-infinity. Here, tlast is the last sampling time at which the concentration is at or above the lower limit of quantification.
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
percentage of AUC0-inf
  Bisoprolol | 3.60 (36.1) | 3.24 (25.5) | 3.83 (21.9) | 3.94 (48.2)
  Amlodipine | 10.9 (40.1) | 10.8 (52.0) | 8.58 (44.7) | 6.81 (64.3)

7. Secondary Outcome: Apparent Terminal Elimination Rate Constant (λz) of Bisoprolol and Amlodipine
Description: λz was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1 per hour
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
1 per hour
  Bisoprolol | 0.0781 (18.1) | 0.0784 (15.4) | 0.0731 (30.2) | 0.0783 (20.6)
  Amlodipine: number analyzed (Participants) | 15 | 13 | 13 | 14
  Amlodipine | 0.0134 (16.1) | 0.0139 (23.5) | 0.0148 (16.5) | 0.0160 (26.1)

8. Secondary Outcome: Apparent Total Body Clearance From Plasma (CL/f) of Bisoprolol and Amlodipine
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
liter per hour
  Bisoprolol | 16.4 (16.6) | 16.4 (21.5) | 17.8 (23.4) | 17.4 (23.2)
  Amlodipine: number analyzed (Participants) | 15 | 13 | 13 | 14
  Amlodipine | 21.3 (34.4) | 23.1 (31.7) | 26.0 (31.4) | 27.4 (34.8)

9. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase Following Extravascular Administration (Vz/f) of Bisoprolol and Amlodipine
Description: Vz/f is defined as the distribution of a study drug between plasma and the rest of the body after oral dosing.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 13 | 14
liter
  Bisoprolol | 209 (17.0) | 209 (15.5) | 243 (31.3) | 223 (19.6)
  Amlodipine: number analyzed (Participants) | 15 | 13 | 13 | 14
  Amlodipine | 1590 (31.0) | 1660 (40.6) | 1750 (30.9) | 1710 (40.5)

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, AEs Leading to Death, and AEs Leading to Discontinuation
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 29
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
Number analyzed (Participants) | 16 | 16 | 14 | 14
Participants
  TEAEs | 0 | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0 | 0
  AEs Leading to Death | 0 | 0 | 0 | 0
  AEs Leading to Discontinuation | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 29
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Fasting: Bisoprolol-Amlodipine FDC | Fasting: Bisoprolol and Amlodipine Separately | Fed: Bisoprolol-Amlodipine FDC | Fed: Bisoprolol and Amlodipine Separately
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT03226275/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT03226275/SAP_001.pdf